CLINICAL TRIAL: NCT01943929
Title: Correlation Between Headaches and Septum and Nasal Mucosa Contact
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Yves Bohrer Costa, MD, Hospital Israelita Albert Einstein
Other Study IDs: IIEP 1392-11
Record Dates: First submitted 2012-12-07; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Nasal Septum Deviation; Headache
Keywords: Nasal septum; Headache; Mucosa contact point headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Headache is the most common complaint to neurologists. In the 80´s and 90's few papers, with limited number of patients, have proposed the association between nasal septum contact and headache. The International Classification of Headaches Disorders proposed specific diagnostic criteria for this entity.

With the major use of CT scans, the contact between nasal mucosa and septum is daily observed in many patients without complaint of headache.

The purpose of this study is to determine if there is any correlation between nasal and septum mucosa contact and the prevalence of headache. The investigators hypothesized that no correlation will be found using CT scans in a large series of patients.

DETAILED DESCRIPTION:
Every patient older than 18 years old whom underwent sinuses or facial computed tomography will be asked to answer a questionnaire, where he will be able to describe his headache features (if present) . This information will be correlated with patient images findings, which are going to be evaluated by head and neck radiologists blinded for clinical information. Logistic regression model will be used to verify this association; the presence of sinusitis and fever will used be as covariates.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years whom underwent sinuses or facial tomography.

Exclusion Criteria:

* Patients with clinical history of trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients older than 18 years whom underwent sinuses or facial tomography.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Complain of Headache during last 3 months (binary response - question answered by the patient at the moment of CT scan) | within less than a day from the date that CT scan is performed
  In order to analyze the effect of nasal mucosal contact points explaining the presence of headache we are going to perform a logistic regression model with the following explanatory variables: grade and location of the contact between nasal septum and nasal mucosa (8 dummy variables) and history of previous nasal surgery. Our hypothesis is that the presence of headache will not be explained by any of these variables. In addition we will also include in this model the following variables: fever, tomographic signs of sinusitis, obliteration of nasal sinus pathways, gender.

CONTACTS AND LOCATIONS:
Overall Officials: Yves B Costa, MD, Principal Investigator — Hospital Israelita Albert Einstein; Ellison F Cardoso, MD, Study Director — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil